CLINICAL TRIAL: NCT05198401
Title: The Impact of the Previous Exposure to Covid-19 Virus Infection on the Outcome of ICSI Cycles
Status: Completed | Type: Observational
Sponsor: Al Baraka Fertility Hospital (Other)
Responsible Party: Principal Investigator, Dr. Kamal Rageh, Doctor, Al Baraka Fertility Hospital
Other Study IDs: covid/kamal
Record Dates: First submitted 2022-01-15; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; IVF
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months

GROUPS / COHORTS (2):
- 1: (previous covid-19 positive) n. =88
  Interventions: Other: covid-19
- 2: (covid-19 negative) n.=91

INTERVENTIONS:
Other: covid-19 — viral infection
  Groups: 1

SUMMARY:
Whilst the global COVID-19 pandemic is still evolving and there are many unknowns about the long-term effects of the virus on fertility and pregnancy, we found ourselves in need to offer some evidence-based guidance, that's why we decided to go for this study, to evaluate the relation of the covid-19 and the outcome of IVF/ICSI cycles. we found that there is no clear evidence that the previous exposure to Covid-19 virus infection can affect the outcome of ICSI cycles significantly.

DETAILED DESCRIPTION:
This is an observational study, for 122 ICSI cycles conducted in Al- Baraka Fertility Hospital, Manama, Bahrain, and Al-Manea hospital, KSA between August 2020 and May 2021, and it was approved by the ethical committees. We compared the outcome results of those patients who got recovered from previous exposure to covid-19 (study group) with results of non-infected comparable patients (control group) After comparison of the basal characteristics in both groups, and we got assured that there is no significant difference regarding the demographic criteria between both groups, we found that there is no significant difference regarding the duration of stimulation, the total dose of stimulation, number of oocytes retrieved, number of metaphase 2 oocytes (MII), number of grade1-2 embryos, number of transferred embryos, day of embryo transfer and fertilization rate.

Although the fertilization rate was higher in Covid-19 free patients (52% vs. 50.6%), however, this difference is not statistically significant.

In the same way, the pregnancy rate was also higher in the covid-19 negative group (45.1% vs. 36.4%); however this difference was not statistically significant.

ELIGIBILITY:
* Inclusion criteria were women who got recovered from Covid-19 based upon their history with positive test results confirmed via BeAware Bahrain phone application and Tawakkalna Saudi phone application; with age below 38 yrs., body mass index (BMI) below 30 kg/m2, who underwent antagonist protocol for IVF
* Exclusion criteria were chromosomal and genetic disorders, age> 38 years, BMI > 30, abnormal ultrasonogram of the uterine cavity (acquired or congenital), those who underwent long agonist protocol, and those cases with severe male factor, and abnormal embryos not suitable for transfer, we excluded also patients with those who got vaccinated against Covid-19 and those with current infection.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: All women underwent individualized antagonist protocol
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-02 (Actual)

PRIMARY OUTCOMES:
number of mature oocytes (MII) | 10 days
  how many mature oocytes

SECONDARY OUTCOMES:
total number of blastocysts | 15 days
  number of blastocysts
B-hcg | 4 weeks
  the clinical pregnancy rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Kamal Eldin Abdalla Rageh, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided